CLINICAL TRIAL: NCT03427697
Title: Effect of Virtual Reality and Accommodation Relax Techniques in Combination on Controlling Myopia Development in School-aged Children
Brief Title: Effect of VR and Accommdation Relax on Controlling Myopia in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Principal Investigator, Shi-Ming Li, Associate professor, Beijing Tongren Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: TRECKY20170704
Record Dates: First submitted 2017-12-17; First posted 2018-02-09 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Myopia; Accommodation Spasm; Children
MeSH Terms: conditions — Myopia; Spasm

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Head-mounted video display which shows video with virtual reality and accommodation relax technique in combination,40 minutes per day
  Interventions: Device: Virtual reality and accommodation relax techniques in combination
- Control group (No Intervention): No intervention will be performed in the control group

INTERVENTIONS:
Device: Virtual reality and accommodation relax techniques in combination — The children will be given head-mounted video display to watch video at break of classes, 40 minutes per day in total. The video will be shown by virtual reality and accommodation relax techniques in combination.
  Arms: Intervention group

SUMMARY:
This study evaluates the effect of virtual reality and accommodation relax technique on controlling onset and development of myopia in school-aged children. Half of the children will receive head-mounted video display which shows video with virtual reality and accommodation relax technique in combination, while the other half will receive no intervention.

ELIGIBILITY:
Inclusion Criteria:

* Best corrected visual acuity >=20/20 for each eye;
* Astigmastism less than 1.5 D;
* Anisometropia less than 1.0D;
* No other ocular or systematic diseases;

Exclusion Criteria:

* Can not endure virtual reality video;
* Can not cooperate with ocular examinations;
* Receiving other interventions for controlling myopia;

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1000 (Estimated)
Dates: Start 2020-09-18 (Estimated); Primary Completion 2022-12-18 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Myopia progression | One year
  The change in spherical equivalent
Axial elongation | One year
  Chnage in axial length

SECONDARY OUTCOMES:
Accommodative lag | One week and One month
  Difference between accommodative demand and accommodative response measured by an open-field autorefractor (WAM-5500, Grand Seiko Co Ltd, Hiroshima, Japan)

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tongren Hospital, Beijing, Beijing Municipality, China